CLINICAL TRIAL: NCT01736384
Title: Can Genetic Changes Predict Weight Loss and Outcome After Bariatric Surgery and Can it Related to Virus Infection and Function of Liver and Adipose Tissue as Well as Lipid and Protein Profiles.
Brief Title: Can Genetic Markers Predict Weight Loss After Gastric By-pass Surgery
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other); Ersta Hospital, Sweden (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Erik Näslund, Professor, Karolinska Institutet
Other Study IDs: 2008/1010-31/3
Record Dates: First submitted 2012-11-12; First posted 2012-11-29 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass; Cholecystectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue biopies, liver and subcutaneous and omental fat Whole blood EDTA-plasma Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obesity: Gastric bypass surgery and non-obese controls undergoing cholecystectomy
  Interventions: Procedure: Gastric bypass or cholecystectomy

INTERVENTIONS:
Procedure: Gastric bypass or cholecystectomy

SUMMARY:
There is a variability in weight loss after gastric bypass surgery for obesity despite a standardised surgical procedure. This study aims to investigate if genetic markers can predict outcome after gastric by-pass surgery in treatment of obesity. The investigators will also study if adenovirus infection can influence the outcome after surgery. In a subgroup of patients, hormonal changes after gastric by-pass surgery will be assessed. Lipid and protein patterns will be assessed in plasma and tissues. Omental and subcutaneous fat as well as liver biopsies and whole blood are stored in a biobank. The same tissues will be collected from non-obese controls undergoing gallbladder surgery.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic gastric by-pass with BMI greater than 35

Exclusion Criteria:

* unable to understand swedish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obesity
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Genetic markers | day of surgery and 1 and 2 years after surgery
  Blood samples and tissue biopsies taken at the time of surgery and at follow-up.

SECONDARY OUTCOMES:
Lipid and protein patterns in plasma and tissues | day of surgery and at 1 and 2 years postoperatively
  Blood samples taken and tissue biopsies taken at the time of surgery and at follow-up
Previous viral infection | At time of surgery
  Blood samples taken before surgery
Genexpression and comorbid disease | At time of bariatric surgery and 1-2 years postoperatively
  Gene expression studies in tissue biopsies and whole blood at time of surgery and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Erik Näslund, Professor, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Karolinska Institutet, Ersta Hospital, Stockholm
  - Karolinska Institutet, Danderyds Hospital, Stockholm
  - Karolinska University Hospital, Stockholm